CLINICAL TRIAL: NCT03305406
Title: Parkdale Infant Nutrition Security Targeted Evaluation Project (PINSTEP): Formative Research (Objective 2-Focus Group & Interview)
Brief Title: Parkdale Infant Nutrition Security Targeted Evaluation Project: Focus Groups & Interviews
Acronym: PINSTEP-2
Status: Completed | Type: Observational
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Daniel Sellen, Professor, University of Toronto
Other Study IDs: 34482-2
Record Dates: First submitted 2017-09-27; First posted 2017-10-10 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Breastfeeding; Breast Pumping; Infant Nutrition; Vulnerable Population
MeSH Terms: conditions — Breast Feeding; Breast Milk Expression | interventions — Focus Groups; Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Focus Group Participants: Semi-structured focus groups
  Interventions: Other: Focus groups
- Interview Participants: One-on-one interviews
  Interventions: Other: Interviews

INTERVENTIONS:
Other: Focus groups — Focus groups will be conducted to gather information on clients view of a community support program focusing on healthy infant nutrition
  Groups: Focus Group Participants
Other: Interviews — Interviews will be conducted to gather information on clients view of a community support program focusing on healthy infant nutrition
  Groups: Interview Participants

SUMMARY:
In Toronto Ontario, the Parkdale Community Health Centre operates a community outreach program entitled Parkdale Parents' Primary Prevention Project (5P's). The 5P's provides weekly pre- and post-natal support and education programs for clients. This includes an infant feeding program for mothers with infants 0-6 months (Feeding Tiny Souls). The 5P's has a diverse client-base; the program is aimed at women who are in challenging life circumstances, therefore, clients may include low-income or single mothers and newcomers to Canada.

The overall goal of this research is to optimize the existing 5P's program. Program acceptability is an essential component of the process evaluation to understand the experiences of mothers and the perceived supports and barriers of the program. Specifically, the aim of this project is twofold: 1) to investigate the perceptions and experiences of accessibility of a postnatal community program and 2) to explore the perceptions of, and attitudes toward, a community infant feeding program offering lactation consultant and breast pump resources. This study will use a qualitative approach by way of semi-structured focus groups and interviews. The study population will consist of women who enrolled in 5P's prenatally and have delivered their infant. This will include women who did and did not continue to participate in the postnatal program and/or Feeding Tiny Souls after delivery. The investigators will specifically seek women who participated in the prenatal program, but did not take part in the postnatal program and/or Feeding Tiny Souls to understand why participants did not access these resources and gather information on their views of these postnatal program components. The hypothesis is that the postnatal community program is a source of support for clients, but that it needs to be expanded to include more clients and the infant feeding program is an important support for helping clients to provide breast milk to their infant.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in Parkdale Parents' Primary Prevention Project (5P's) prenatally
* Delivered their infant between June 1, 2016 and August 16, 2017

Exclusion Criteria:

* Unavailable to participate in a focus group or interview
* Only attended Parkdale Parents' Primary Prevention Project (5P's) postnatally

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Clients enrolled in the Parkdale Parents' Primary Prevention Project (5P's) at the Parkdale Community Health Centre in Toronto, Ontario, Canada
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2017-08-18 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
Perceptions of, and attitudes toward, a community infant feeding program offering lactation consultant and breast pump resources as assessed by group responses to targeted probes during postnatal focus groups and interviews | 60 minutes (participants are 1-14 months postpartum)
  Qualitative summary of perceptions and attitudes regarding a community infant feeding program

SECONDARY OUTCOMES:
Perceptions and experiences of accessibility of a postnatal community program as assessed by group responses to targeted probes during postnatal focus groups and interviews | 60 minutes (participants are 1-14 months postpartum)
  Qualitative summary of perceptions and experiences of accessibility regarding a community infant feeding program

CONTACTS AND LOCATIONS:
Overall Officials: Jane Francis, MSc, Principal Investigator — University of Toronto
Locations (1):
- Parkdale Community Health Centre, Toronto, Ontario, Canada

REFERENCES:
- [Result] Francis J, Mildon A, Stewart S, Underhill B, Tarasuk V, Di Ruggiero E, Sellen D, O'Connor DL. Vulnerable mothers' experiences breastfeeding with an enhanced community lactation support program. Matern Child Nutr. 2020 Jul;16(3):e12957. doi: 10.1111/mcn.12957. Epub 2020 Jan 26. PMID 31984642